CLINICAL TRIAL: NCT03074253
Title: Cardiovascular Imaging and Biomarker Analyses (CIBER)
Acronym: CIBER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Michael Behnes, Dr. med, Universitätsmedizin Mannheim
Other Study IDs: 2014-615N-MA
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease; Heart Diseases; Heart Failure
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Heart Failure | interventions — Echocardiography; Magnetic Resonance Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One peripheral blood withdraws in EDTA, citrate, ammonium heparin, serum tubes within 24 hours before cardiac imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Patients are undergoing echocardiography
Diagnostic Test: magnetic resonance imaging — Patients are undergoing magnetic resonance imaging
  Other Names: MRI
Diagnostic Test: computed tomography — Patients are undergoing computed tomography
  Other Names: CT
Diagnostic Test: blood withdrawl — Peripheral blood samples are being collected from all patients

SUMMARY:
"Cardiovascular Imaging and Biomarker Analyses (CIBER)" is a single-center, prospective and observational study evaluating the expression of novel biomarkers in patients undergoing cardiacvascular imaging within clinical routine care. It is aimed to evaluate associations with biomarker expressions with ascertained cardiac imaging parameters.

DETAILED DESCRIPTION:
"Cardiovascular Imaging and Biomarker Analyses (CIBER)" is a single-center, prospective and observational study evaluating the expression of novel biomarkers in patients undergoing cardiacvascular imaging within clinical routine care. It is aimed to evaluate associations with biomarker expressions with ascertained cardiac imaging parameters. Furthermore the prognostic value of biomarkers and imaging parameters on mid-term and long-term prognosis will be evaluated. Novel biomarkers will comprise blood derived biomarkers including neurohormones, proteins, cytokines, microRNAs and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* patients with low to intermediate risk for coronary artery disease

Exclusion Criteria:

* under 18 years
* mechanical heart valve
* pulmonary embolism
* deep vein thrombosis
* myocardial infarction within the last 3 months
* electrical cardioversion within 30 days
* status after heart transplant
* transient ischemic attack (TIA) or stroke within last 30 days
* intracerebral bleeding within the last 2 months
* acute infection
* existing or planned pregnancy
* chronic kidney disease with eGFR < 40 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac imaging (i.g. echocardiography, cardiac MRI, cardiac CT) within the clinical routine.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-12-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker levels before cardiac imaging | 24 hours before cardiac imaging

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Akin, Prof. Dr., Study Director — University Medical Center Mannheim
Locations (1):
- First Department of Medicine, University Medical Centre Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SH, Behnes M, Natale M, Hoffmann J, Reckord N, Hoffmann U, Budjan J, Henzler T, Papavassiliu T, Borggrefe M, Bertsch T, Akin I. Galectin-3 Reflects Mitral Annular Plane Systolic Excursion Being Assessed by Cardiovascular Magnetic Resonance Imaging. Dis Markers. 2016;2016:7402784. doi: 10.1155/2016/7402784. Epub 2016 Dec 1. PMID 28044067
- [Background] Behnes M, Lang S, Breithardt OA, Kaden JJ, Haghi D, Ahmad-Nejad P, Elmas E, Wolpert C, Borggrefe M, Neumaier M, Brueckmann M. Association of NT-proBNP with severity of heart valve disease in a medical patient population presenting with acute dyspnea or peripheral edema. J Heart Valve Dis. 2008 Sep;17(5):557-65. PMID 18980090
- [Background] Behnes M, Bertsch T, Weiss C, Ahmad-Nejad P, Akin I, Fastner C, El-Battrawy I, Lang S, Neumaier M, Borggrefe M, Hoffmann U. Triple head-to-head comparison of fibrotic biomarkers galectin-3, osteopontin and gremlin-1 for long-term prognosis in suspected and proven acute heart failure patients. Int J Cardiol. 2016 Jan 15;203:398-406. doi: 10.1016/j.ijcard.2015.10.127. Epub 2015 Oct 20. PMID 26539964
- [Background] Behnes M, Brueckmann M, Lang S, Espeter F, Weiss C, Neumaier M, Ahmad-Nejad P, Borggrefe M, Hoffmann U. Diagnostic and prognostic value of osteopontin in patients with acute congestive heart failure. Eur J Heart Fail. 2013 Dec;15(12):1390-400. doi: 10.1093/eurjhf/hft112. Epub 2013 Jul 12. PMID 23851388
- [Derived] Ansari U, Behnes M, Hoffmann J, Weidner K, Kuche P, Rusnak J, Kim SH, Natale M, Reckord N, Lang S, Hoffmann U, Bertsch T, Fatar M, Borggrefe M, Akin I. Galectin-3 reflects the echocardiographic quantification of right ventricular failure. Scand Cardiovasc J. 2021 Dec;55(6):362-370. doi: 10.1080/14017431.2021.1995036. Epub 2021 Nov 5. PMID 34738853
- [Derived] Hoffmann J, Behnes M, Ansari U, Weidner K, Kuche P, Rusnak J, Kim SH, Natale M, Reckord N, Lang S, Hoffmann U, Bertsch T, Fatar M, Borggrefe M, Akin I. The association of high-sensitivity cardiac troponin I and T with echocardiographic stages of heart failure with preserved ejection fraction. Ann Clin Biochem. 2019 Jul;56(4):431-441. doi: 10.1177/0004563219841644. Epub 2019 May 21. No abstract available. PMID 31112389
- [Derived] Rusnak J, Behnes M, Henzler T, Reckord N, Vogler N, Meyer M, Hoffmann U, Natale M, Hoffmann J, Hamed S, Weidner K, Lang S, Mukherji A, Haubenreisser H, Schoenberg SO, Borggrefe M, Bertsch T, Akin I. Comparative analysis of high-sensitivity cardiac troponin I and T for their association with coronary computed tomography-assessed calcium scoring represented by the Agatston score. Eur J Med Res. 2017 Nov 16;22(1):47. doi: 10.1186/s40001-017-0290-9. PMID 29145895
- [Derived] Rusnak J, Behnes M, Reckord N, Hoffmann U, Natale M, Hoffmann J, Weidner K, Lang S, Mukherji A, Kruska M, Henzler T, Schoenberg SO, Borggrefe M, Bertsch T, Akin I. High Sensitivity Troponins Discriminate Different Morphologies of Coronary Artery Plaques Being Assessed by Coronary Computed Tomography Angiography. Dis Markers. 2017;2017:9306409. doi: 10.1155/2017/9306409. Epub 2017 Jul 18. PMID 28804199